CLINICAL TRIAL: NCT04710602
Title: A Prospective Follow-up of Patients Treated With Muscle Sparing, Minimally Invasive Open Surgical Technique for Unstable Chest Wall After Trauma
Brief Title: Prospective Follow up of Minimally Invasive Chest Wall Surgery After Trauma
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Erik Öberg Westin, Principal Investigator, Sahlgrenska University Hospital
Other Study IDs: FoU-274457
Record Dates: First submitted 2020-12-18; First posted 2021-01-14 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Rib; Fracture, Multiple, With Flail Chest
Keywords: Chest wall; Trauma; Minimally invasive; Surgery; Muscle sparing
MeSH Terms: conditions — Fractures, Bone; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Minimally invasive: Patients who underwent surgery with a muscle sparing, minimally invasive technique for unstable chest wall after trauma.
  Interventions: Procedure: Minimally invasive surgical fixation of unstable rib cage
- Historical control: Patients who underwent surgery with large incisions and simultaneous thoracotomy for unstable chest wall after trauma.
  Interventions: Procedure: Large incision surgical fixation of unstable rib cage.

INTERVENTIONS:
Procedure: Minimally invasive surgical fixation of unstable rib cage — Minimally invasive and muscle sparing surgical fixation of ribs and/or sternum in an unstable segment of the chest wall (flail chest) with titan plates or medullary nails (MatrixRib Fixation System, DepuySynthes).
  Groups: Minimally invasive
Procedure: Large incision surgical fixation of unstable rib cage. — Surgical fixation of ribs and/or sternum in an unstable segment of the chest wall (flail chest) with titan plates or medullary nails (MatrixRib Fixation System, DepuySynthes). Large non muscle sparing incision with simultaneous thoracotomy.
  Groups: Historical control

SUMMARY:
The purpose of this study is to assess the outcome of a muscle sparing, minimally invasive open surgical technique for unstable ribcage injuries after trauma. The investigators will compare the results from the study participants to a historical cohort who were operated with a different surgical technique with large incisions and simultaneous thoracotomy.

DETAILED DESCRIPTION:
This is a prospective follow-up study where the investigators aim to study patients who have undergone surgery with a muscle sparing, minimally invasive technique for unstable ribcage after trauma. The investigators plan on seeing the participants as out patients 6 months and 1 year after surgery. The results will be compared to results from a historical cohort with patients who participated in earlier studies with a different surgical method with large incisions and simultaneous thoracotomy. The investigators plan on including 50 patients since a preliminary analysis has suggested this should be enough to notice statistically significant differences between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chest wall trauma who underwent surgical stabilisation for unstable chest wall using a minimally invasive, muscle sparing technique without thoracotomy or thoracoscopy no more than 6 months prior to inclusion.

Exclusion Criteria:

* Severe head injury (Abbreviated Injury score (AIS) >3)
* Spinal injury
* Neurological or musculoskeletal disease affecting chest wall mobility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients surgically treated at our trauma ward for unstable chest wall due to trauma. Consecutive sampling.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Vital capacity of the lungs. | One year after surgery.
  Vital capacity (VC) measured with spirometry.
Forced vital capacity of the lungs. | One year after surgery.
  Forced vital capacity (VC) measured with spirometry.
Forced expiratory volume of the lungs. | One year after surgery.
  Forced expiratory volume in 1 second (FEV1) measured with spirometry.
Forced expiratory volume percent of the lungs. | One year after surgery.
  Forced expiratory volume in 1 second divided with forced vital capacity, measured with spirometry.
Peak expiratory flow of the lungs. | One year after surgery.
  Peak expiratory flow measured with spirometry.

SECONDARY OUTCOMES:
Disability | Six months and one year after surgery.
  Degree of disability assessed with Disability Rating Index (DRI) scale ranging from 0-100 where higher scores indicate more disability.
Physical activity | Six months and one year after surgery.
  Physical activity assessed with Grimby activity scale ranging from 1-6 where 6 indicates the highest level of activity.
Shoulder mobility | Six months and one year after surgery.
  Shoulder mobility assessed with Boström index, a scale ranging from 5-30 for each shoulder where 30 represents the greatest range of movement.
Respiratory movement | Six months and one year after surgery.
  Movement of chest wall during respiration measured with Respiratory Movement Measuring Instrument (RMMI).
Strength of respiratory muscles | Six months and one year after surgery.
  Strength of respiratory muscles measured with Maximal Inspiratory Pressure (MIP) and Maximal Expiratory Pressure (MEP).
Quality of life EQ-5D-5L | Six months and one year after surgery.
  Quality of life assessed with the EuroQol (European Quality of Life) Five Dimension Five Level Scale (EQ-5D-5L). A 5-dimensional scale in which each dimension has 5 levels where 1 represents the best outcome and 5 represents the worst outcome.
Radiological healing | One year after surgery.
  Radiological signs of healing of the participants rib fractures assessed with CT scan. Fractures will be denoted as healed, partially healed or with no signs of healing.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Westin, MD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No
Sharing data with other researchers will be considered by request.

REFERENCES:
- [Background] Bemelman M, van Baal M, Yuan JZ, Leenen L. The Role of Minimally Invasive Plate Osteosynthesis in Rib Fixation: A Review. Korean J Thorac Cardiovasc Surg. 2016 Feb;49(1):1-8. doi: 10.5090/kjtcs.2016.49.1.1. Epub 2016 Feb 5. PMID 26889439
- [Background] Caragounis EC, Fagevik Olsen M, Pazooki D, Granhed H. Surgical treatment of multiple rib fractures and flail chest in trauma: a one-year follow-up study. World J Emerg Surg. 2016 Jun 14;11:27. doi: 10.1186/s13017-016-0085-2. eCollection 2016. PMID 27307787
- [Background] Granetzny A, Abd El-Aal M, Emam E, Shalaby A, Boseila A. Surgical versus conservative treatment of flail chest. Evaluation of the pulmonary status. Interact Cardiovasc Thorac Surg. 2005 Dec;4(6):583-7. doi: 10.1510/icvts.2005.111807. Epub 2005 Sep 15. PMID 17670487
- [Background] Granhed HP, Pazooki D. A feasibility study of 60 consecutive patients operated for unstable thoracic cage. J Trauma Manag Outcomes. 2014 Dec 30;8(1):20. doi: 10.1186/s13032-014-0020-z. eCollection 2014. PMID 25642282
- [Background] Marasco SF, Davies AR, Cooper J, Varma D, Bennett V, Nevill R, Lee G, Bailey M, Fitzgerald M. Prospective randomized controlled trial of operative rib fixation in traumatic flail chest. J Am Coll Surg. 2013 May;216(5):924-32. doi: 10.1016/j.jamcollsurg.2012.12.024. Epub 2013 Feb 13. PMID 23415550
- [Background] Tanaka H, Yukioka T, Yamaguti Y, Shimizu S, Goto H, Matsuda H, Shimazaki S. Surgical stabilization of internal pneumatic stabilization? A prospective randomized study of management of severe flail chest patients. J Trauma. 2002 Apr;52(4):727-32; discussion 732. doi: 10.1097/00005373-200204000-00020. PMID 11956391
- [Derived] Westin EO, Olsen MF, Caragounis EC. Comparison of long-term outcome between muscle sparing and non-muscle sparing surgical techniques in rib plating. Eur J Trauma Emerg Surg. 2025 May 20;51(1):212. doi: 10.1007/s00068-025-02881-z. PMID 40392360